CLINICAL TRIAL: NCT00638001
Title: Impact of Conservative Treatment by Custom-made Orthoses in Patients With Haemophilic Ankle Arthropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: READ-LOBET-01
Record Dates: First submitted 2008-02-26; First posted 2008-03-18 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Haemophilia A; Haemophilia B
Keywords: patients with haemophilia A moderate or severe; patients with haemophilia B moderate or severe
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: custom-molded insoles and custom-molded shoes — * custom-made insoles in "PELITE" foam (hypoallergenic prosthesis grade foam) or leather top cover cork insoles for patients suffering of mild to moderate ankle arthropathy
  * custom-molded shoes in leather for patients suffering of end-stage ankle arthropathy

SUMMARY:
The purpose of this study intend to evaluate the effectiveness of functional orthoses (including custom-made insoles and shoes) for preventing and controlling repetitive haemarthrosis in patients suffering of haemophilic ankle arthropathy, as well as the orthoses' impact on foot health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* haemophilia A or B, aged more than 13 years

Exclusion Criteria:

* impossibility to walk on a treadmill
* recent joint haemarthrosis or muscle haematoma

Ages: 13 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Gait analysis, foot pressure measurement, specific joint score | To, T1 (3months) and T2 (6months)

CONTACTS AND LOCATIONS:
Locations (1):
- cliniques Universitaires Saint Luc, Brussels, Belgium